CLINICAL TRIAL: NCT03733314
Title: Early Phase 2 Clinical Trial of E6011 in Patients With Active Crohn's Disease
Brief Title: A Study of E6011 in Participants With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E6011-ET2; 2018-002109-70 (EudraCT Number); 184139 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; E6011; Inflammatory Bowel Diseases; Gastroenteritis; Gastrointestinal tract
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Gastroenteritis | interventions — quetmolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E6011 (Experimental)
  Interventions: Drug: E6011
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6011 — E6011, infusion, intravenously.
  Arms: E6011
Drug: Placebo — Placebo, infusion, intravenously.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to examine the efficacy and safety of E6011 at 12 weeks after administration by means of double-blind placebo-controlled trial.

DETAILED DESCRIPTION:
Participants with moderate to severe Crohn's disease will be enrolled in this study.

The study will include screening period, remission-induction period (double-blind), rescue period (open-label), extension period (open-label), post-observation period, and a follow-up period.

At the end of remission-induction period, participants with reduction in Crohn's disease activity index (CDAI) score of 70 points or more when compared to baseline will move on to the open-label extension period, and participants with less than 70 points reduction in CDAI score will move on to the rescue period. At the end of the rescue period, participants with a reduction in the CDAI of 70 points or more will move on to the open-label extension period and with less than 70 points reduction in the CDAI score will be discontinued.

The post-observation period will include in-person assessment after the completion or discontinuation of the extension period, and participants will be contacted by telephone, etc. after the last dose of study drug administration. Participants will be contacted over phone after the last dose of study drug administration for follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Has diagnosed on basis of clinical findings, endoscopic findings, etc. with small intestine-type, small and large-intestine type, or large-intestine type Crohn's disease at least 12 weeks before giving consent.
2. With a baseline (at week 0 before the start of investigational medicinal product [IMP] administration) disease severity ranging from moderate to severe. CDAI score between 220 and 450, and a PRO2 score between 14 and 34.
3. With a SES-CD >=7 (or for participants with isolated ileal disease, >=4 in ileum segment) in the screening period, with one or more ulcers (in SES-CD score, ulcer presence subscore >=1 in any segment) assessed by colonoscopy and confirmed by a centralised review.
4. Who received adrenocorticosteroids or immunomodulators in the past, but showed no therapeutic response (insufficient response) or the drugs were not tolerated (intolerance). Alternatively, participants who cannot taper adrenocorticosteroids (dependence). Alternatively, participants who showed no therapeutic response after administering biologic(s) (primary nonresponse), participants who initially showed therapeutic response but it lessened or disappeared afterwards (secondary nonresponse), or participants who did not tolerate the drug (intolerance).
5. If the participants are taking aminosalicylic acid (5-ASA), salazosulfapyridine, or antibiotics for the treatment of Crohn's disease (metronidazole, ciprofloxacin, etc.), the dosage and administration have not changed for at least 4 weeks prior to the start of the IMP administration.
6. If the participants are taking under 30 milligram per day (mg/day) of oral prednisolone (or equivalent adrenocorticosteroid) or 9 mg/day or less of oral budesonide, the dosage and administration have not changed for at least 4 weeks prior to the start of the IMP administration.
7. If the participants are taking azathioprine (AZP), 6-mercaptopurine (6-MP) or methotrexate (MTX), the dosage and administration have not changed for at least 8 weeks prior to the start of the IMP administration.

Exclusion Criteria:

1. Diagnosed with ulcerative colitis or indeterminate colitis.
2. Diagnosed with gastrointestinal epithelial dysplasia.
3. Who have an abscess or are suspected to have one.
4. With an artificial anus, ileo-anal pouch or fistula.
5. With symptomatic or high-grade gastrointestinal stenosis (participants who require expansion by endoscopy or who require have SES-CD score stenosis sub-score of 3, etc.).
6. Who, after undergoing small bowel resection, have been diagnosed with a short bowel syndrome, which makes maintaining caloric intake difficult.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2024-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- 49, CCR Ostrava, s.r.o, Ostrava, Czechia
- Hungary (2):
  - 15, University of Debrecen Clinical Centre, Debrecen
  - 19, Semmelweis university, Győr
- Japan (34):
  - 4, Nagoya, Aichi-ken
  - 17, Toyota, Aichi-ken
  - 10, Abiko, Chiba
  - 31, Kashiwa, Chiba
  - 27, Kitakyushu, Fukuoka
  - 39, Kitakyushu, Fukuoka
  - 29, Kasamatsuchō, Gifu
  - 41, Kure, Hiroshima
  - 38, Asahikawa, Hokkaido
  - 26, Sapporo, Hokkaido
  - 37, Kobe, Hyōgo
  - 7, Nishinomiya, Hyōgo
  - 32, Kanazawa, Ishikawa-ken
  - 8, Takamatsu, Kagawa-ken
  - 52, Isehara, Kanagawa
  - 30, Ōiso, Kanagawa
  - 28, Urasoe, Okinawa
  - 42, Hirakata, Osaka
  - 51, Hamamatsu, Shizuoka
  - 50, Shuntougun, Shizuoka
  - 2, Bunkyo, Tokyo
  - 33, Hachiōji, Tokyo
  - 34, Kodaira, Tokyo
  - 3, Minato, Tokyo
  - 6, Mitaka, Tokyo
  - 43, Shinagawa-Ku, Tokyo
  - 1, Shinjuku, Tokyo
  - 36, Akita
  - 25, Fukuoka
  - 35, Fukuoka
  - 11, Gifu
  - 5, Kagoshima
  - 40, Kanazawa
  - 24, Osaka
- Poland (4):
  - 21, Vitamed Galaj i Cichomski sp.j., Bydgoszcz
  - 22, Vita Longa, Katowice
  - 20, Clinical Research Center sp. z o.o., Medic-R Sp. k., Poznan
  - 23, Centrum Badań Klinicznych - Ośrodek Badań Wczesnej Fazy, Wroclaw
- Russia (5):
  - 45, Federal Siberian Research and Clinical Center, Krasnoyarsk
  - 44, LLC, Novosibirskiy Gastrocenter, Novosibirsk
  - 46, Pyatigorsk City Clinical Hospital, Pyatigorsk
  - 48, LLC Clinic, UZI 4D, Pyatigorsk
  - 47, City Hospital of Saint Martyr Elizaveth, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 49 investigative sites in Japan, Czech Republic, Hungary, Poland, and Russia from 25 April 2019 to 03 April 2024.
Pre-assignment Details: A total of 65 participants were screened, of which 40 were screen failures and 25 were enrolled to receive study treatment.
Groups:
- E6011 10 mg/kg: Participants with moderate to severe active Crohn's disease received E6011 10 milligram per kilogram (mg/kg), intravenous (IV) infusion once, at Weeks 0, 1, 2 then every 2 weeks up Week 10 during the Remission Induction Period, thereafter, non-responder participants continued E6011 treatment at Weeks 12, 13, 14 then every 2 weeks up to Week 22 during the Rescue Period. Responder participants at Week 12 continued E6011 treatment, every 4 weeks from Week 12 to Week 48 and responders at Week 24 continued E6011 treatment, every 4 weeks, from Week 24 to Week 60 during the Extension Period.
- Placebo Then E6011 10 mg/kg: Participants with moderate to severe active Crohn's disease received placebo, IV infusion once, at Weeks 0, 1, 2 then every 2 weeks up Week 10 during the Remission Induction Period, thereafter, non-responder participants received E6011 10 mg/kg, IV infusion once, at Weeks 12, 13, 14 then every 2 weeks up to Week 22 during the Rescue Period. Responder participants at Week 12 continued E6011 treatment, every 4 weeks from Week 12 to Week 48 and responders at Week 24 continued E6011 treatment, every 4 weeks, from Week 24 to Week 60 during the Extension Period.
Period: Remission-induction Period: (Weeks 0-12)
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Started | 12 | 13
CDAI Responders at Week 12 | 5 | 6
CDAI Non-responders at Week 12 | 5 | 7
Completed | 10 | 13
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Rescue Period: (Weeks 12 to 24)
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Started (Participants with a reduction in the Crohn's Disease Activity Index (CDAI) of less than 70 compared to baseline (non-responders) after finishing evaluation in Week 12 of the remission-induction period were transferred to the rescue period. The rescue period total duration was 12 weeks (from Week 12 to 24).) | 5 | 7
CDAI Responders at Week 24 | 2 | 2
CDAI Non-responders at Week 24 (Participants whose Crohn's Disease Activity Index (CDAI) had not improved by Week 24 were discontinued and were moved on to Post-observation Period.) | 2 | 1
Completed | 4 | 3
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Progressive disease | 0 | 2
Period: Extension Period:(Week 12-52/Week 24-64)
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Started (Participants who finished evaluation at Week 12 of the remission-induction period and who had a CDAI response of 70 or more, and participants who moved on to the rescue period and finished evaluation at Week 24 with a CDAI response of 70 or more were transferred to extension period. The extension period total duration was 40 weeks (i.e., from Weeks 12 to 52 for participants with response at Week 12; and from Weeks 24 to 64 for participants with response at Week 24).) | 7 | 8
Completed | 2 | 5
Not Completed | 5 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Progressive Disease | 1 | 0
Not completed — Other | 3 | 2
Period: Post-observation Period
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Started (All participants who completed or discontinued any of the periods (remission-induction period, rescue period, extension period) were followed up for up to 70 days in post-observation period.) | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included participants to whom the investigational medicinal product (IMP) has been administered after randomization, and who had 1 or more evaluable, post-IMP administration primary efficacy endpoint (that is, to have an evaluable CDAI value at baseline and any other post baseline).
Groups:
- Total: Total of all reporting groups
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (8.7) | 33.2 (12.0) | 31.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response (CR) 100 (CR100) at Week 12
Description: CR100 was defined as clinical response with a reduction of greater than or equal to (>=) 100 points in CDAI score from baseline. The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. The sub scores of abdominal pain (0-3), general well-being (0-4, higher values mean worse well-being), and number of very soft or liquid stools were then summed. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: At Week 12
Population: The FAS included participants to whom the IMP has been administered after randomization, and who had 1 or more evaluable, post-IMP administration primary efficacy endpoint (that is, to have an evaluable (CDAI) value at baseline and any other post baseline).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percentage of participants | 33.3 [9.9 to 65.1] | 23.1 [5.0 to 53.8]
Statistical Analysis 1: Comparison: E6011 10 mg/kg vs Placebo Then E6011 10 mg/kg; Test type: Superiority; Difference = 10.3, 95% CI 2-sided [-24.9 to 45.4] — The difference of percentage was calculated as E6011 minus placebo

2. Secondary Outcome: Percentage of Participants With CR70 and CR100
Description: CR70 was defined as CR with a reduction of >=70 points in CDAI score from baseline. CR100 was defined as clinical response with a reduction of >=100 points in CDAI score from baseline. The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. The sub scores of abdominal pain (0-3), general well-being (0-4, higher values mean worse well-being), and number of very soft or liquid stools were then summed. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: At Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: FAS was used for analysis. Here "number analyzed" ('n') = participants who were evaluable for outcome measure at given time points. As planned, combined data for all the periods (remission-induction, rescue and extension periods) was collected and reported in outcome measure due to same dosing of E6011. From Week 14-24, participants data analyzed simultaneously for rescue and extension period and reported collectively.
Measure: Number; unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percentage of participants
  CR70: Week 2 | 16.7 | 23.1
  CR70: Week 4: number analyzed (Participants) | 11 | 13
  CR70: Week 4 | 45.5 | 23.1
  CR70: Week 8: number analyzed (Participants) | 10 | 13
  CR70: Week 8 | 50.0 | 38.5
  CR70: Week 12: number analyzed (Participants) | 10 | 13
  CR70: Week 12 | 50.0 | 46.2
  CR70: Week 14: number analyzed (Participants) | 4 | 6
  CR70: Week 14 | 25.0 | 33.3
  CR70: Week 16: number analyzed (Participants) | 10 | 10
  CR70: Week 16 | 70.0 | 60.0
  CR70: Week 20: number analyzed (Participants) | 9 | 8
  CR70: Week 20 | 66.7 | 62.5
  CR70: Week 24: number analyzed (Participants) | 8 | 7
  CR70: Week 24 | 62.5 | 71.4
  CR70: Week 28: number analyzed (Participants) | 4 | 7
  CR70: Week 28 | 100.0 | 85.7
  CR70: Week 32: number analyzed (Participants) | 4 | 6
  CR70: Week 32 | 50.0 | 83.3
  CR70: Week 36: number analyzed (Participants) | 4 | 6
  CR70: Week 36 | 100.0 | 83.3
  CR70: Week 40: number analyzed (Participants) | 3 | 4
  CR70: Week 40 | 100.0 | 75.0
  CR70: Week 44: number analyzed (Participants) | 3 | 5
  CR70: Week 44 | 100.0 | 80.0
  CR70: Week 48: number analyzed (Participants) | 3 | 4
  CR70: Week 48 | 66.7 | 100.0
  CR70: Week 52: number analyzed (Participants) | 3 | 3
  CR70: Week 52 | 66.7 | 66.7
  CR70: Week 56: number analyzed (Participants) | 0 | 1
  CR70: Week 56 |  | 100.0
  CR70: Week 60: number analyzed (Participants) | 0 | 2
  CR70: Week 60 |  | 100.0
  CR70: Week 64: number analyzed (Participants) | 0 | 1
  CR70: Week 64 |  | 100.0
  CR100: Week 2 | 16.7 | 15.4
  CR100: Week 4: number analyzed (Participants) | 11 | 13
  CR100: Week 4 | 18.2 | 23.1
  CR100: Week 8: number analyzed (Participants) | 10 | 13
  CR100: Week 8 | 30.0 | 30.8
  CR100: Week 12: number analyzed (Participants) | 10 | 13
  CR100: Week 12 | 40.0 | 23.1
  CR100: Week 14: number analyzed (Participants) | 4 | 6
  CR100: Week 14 | 25.0 | 33.3
  CR100: Week 16: number analyzed (Participants) | 10 | 10
  CR100: Week 16 | 70.0 | 50.0
  CR100: Week 20: number analyzed (Participants) | 9 | 8
  CR100: Week 20 | 55.6 | 50.0
  CR100: Week 24: number analyzed (Participants) | 8 | 7
  CR100: Week 24 | 50.0 | 57.1
  CR100: Week 28: number analyzed (Participants) | 4 | 7
  CR100: Week 28 | 100.0 | 71.4
  CR100: Week 32: number analyzed (Participants) | 4 | 6
  CR100: Week 32 | 50.0 | 83.3
  CR100: Week 36: number analyzed (Participants) | 4 | 6
  CR100: Week 36 | 75.0 | 50.0
  CR100: Week 40: number analyzed (Participants) | 3 | 4
  CR100: Week 40 | 100.0 | 75.0
  CR100: Week 44: number analyzed (Participants) | 3 | 5
  CR100: Week 44 | 66.7 | 80.0
  CR100: Week 48: number analyzed (Participants) | 3 | 4
  CR100: Week 48 | 66.7 | 75.0
  CR100: Week 52: number analyzed (Participants) | 3 | 3
  CR100: Week 52 | 66.7 | 66.7
  CR100: Week 56: number analyzed (Participants) | 0 | 1
  CR100: Week 56 |  | 100.0
  CR100: Week 60: number analyzed (Participants) | 0 | 2
  CR100: Week 60 |  | 50.0
  CR100: Week 64: number analyzed (Participants) | 0 | 1
  CR100: Week 64 |  | 100.0

3. Secondary Outcome: Percentage of Participants With Below 150 CDAI Points
Description: CDAI remission was defined as CDAI score below (<) 150 points. The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. The sub scores of abdominal pain (0-3), general well-being (0-4, higher values mean worse well-being), and number of very soft or liquid stools were then summed. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: At Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: FAS was used for analysis. Here, number analyzed "n"= participants who were evaluable for outcome measure at given time points. As planned, combined data for all the periods (remission-induction, rescue and extension periods) was collected and reported in outcome measure due to same dosing of E6011. From Week 14-24, participants data analyzed simultaneously for rescue and extension period and reported collectively.
Measure: Number; unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percentage of participants
  CDAI <150 points: Week 2 | 0.0 | 7.7
  CDAI <150 points: Week 4: number analyzed (Participants) | 11 | 13
  CDAI <150 points: Week 4 | 0.0 | 15.4
  CDAI <150 points: Week 8: number analyzed (Participants) | 10 | 13
  CDAI <150 points: Week 8 | 20.0 | 30.8
  CDAI <150 points: Week 12: number analyzed (Participants) | 10 | 13
  CDAI <150 points: Week 12 | 10.0 | 15.4
  CDAI <150 points: Week 14: number analyzed (Participants) | 4 | 6
  CDAI <150 points: Week 14 | 0.0 | 16.7
  CDAI <150 points: Week 16: number analyzed (Participants) | 10 | 10
  CDAI <150 points: Week 16 | 20.0 | 30.0
  CDAI <150 points: Week 20: number analyzed (Participants) | 9 | 8
  CDAI <150 points: Week 20 | 11.1 | 37.5
  CDAI <150 points: Week 24: number analyzed (Participants) | 8 | 7
  CDAI <150 points: Week 24 | 12.5 | 42.9
  CDAI <150 points: Week 28: number analyzed (Participants) | 4 | 7
  CDAI <150 points: Week 28 | 100.0 | 42.9
  CDAI <150 points: Week 32: number analyzed (Participants) | 4 | 6
  CDAI <150 points: Week 32 | 50.0 | 83.3
  CDAI <150 points: Week 36: number analyzed (Participants) | 4 | 6
  CDAI <150 points: Week 36 | 25.0 | 33.3
  CDAI <150 points: Week 40: number analyzed (Participants) | 3 | 4
  CDAI <150 points: Week 40 | 66.7 | 50.0
  CDAI <150 points: Week 44: number analyzed (Participants) | 3 | 5
  CDAI <150 points: Week 44 | 33.3 | 60.0
  CDAI <150 points: Week 48: number analyzed (Participants) | 3 | 4
  CDAI <150 points: Week 48 | 0.0 | 50.0
  CDAI <150 points: Week 52: number analyzed (Participants) | 3 | 3
  CDAI <150 points: Week 52 | 33.3 | 66.7
  CDAI <150 points: Week 56: number analyzed (Participants) | 0 | 1
  CDAI <150 points: Week 56 |  | 100.0
  CDAI <150 points: Week 60: number analyzed (Participants) | 0 | 2
  CDAI <150 points: Week 60 |  | 50.0
  CDAI <150 points: Week 64: number analyzed (Participants) | 0 | 1
  CDAI <150 points: Week 64 |  | 100.0

4. Secondary Outcome: Percentage of Participants With at Least 5-point and 8-point Reduction From Baseline in Patient Reported Outcome 2 (PRO2)
Description: Patient reported outcome 2-clinical response 5 (PRO2-CR5) was defined as CR with a reduction of 5 or more points in PRO2 score from baseline. Patient reported outcome 2-clinical response 8 (PRO2-CR8) was defined as CR with a reduction of 8 or more points in PRO2 score from baseline. The PRO2 scale is a patient-reported outcome measure specifically used to assess the severity of Crohn's disease. It is derived from the CDAI and focuses on two main symptoms: abdominal pain and stool frequency. Participants rate their abdominal pain on a scale from 0 (none) to 3 (severe) and report the number of soft or liquid stools they have per day, which are then multiplied by a factor of 2 and 5, respectively. The scores from these two components are combined to give an overall PRO2 score ranging from 0 to no upper limit, with a higher score=worse outcome.
Time Frame: At Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: FAS was used for analysis. Here, "n" = participants who were evaluable for outcome measure at given time points. As planned, combined data for all the periods (remission-induction, rescue and extension periods) was collected and reported in outcome measure due to same dosing of E6011. From Week 14-24, participants data analyzed simultaneously for rescue and extension period and reported collectively.
Measure: Number; unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percentage of participants
  >=5-point reduction: Week 2 | 25.0 | 38.5
  >=5-point reduction: Week 4: number analyzed (Participants) | 11 | 13
  >=5-point reduction: Week 4 | 45.5 | 38.5
  >=5-point reduction: Week 8: number analyzed (Participants) | 10 | 13
  >=5-point reduction: Week 8 | 60.0 | 53.8
  >=5-point reduction: Week 12: number analyzed (Participants) | 10 | 13
  >=5-point reduction: Week 12 | 50.0 | 53.8
  >=5-point reduction: Week 14: number analyzed (Participants) | 4 | 6
  >=5-point reduction: Week 14 | 25.0 | 50.0
  >=5-point reduction: Week 16: number analyzed (Participants) | 10 | 10
  >=5-point reduction: Week 16 | 70.0 | 60.0
  >=5-point reduction: Week 20: number analyzed (Participants) | 9 | 8
  >=5-point reduction: Week 20 | 77.8 | 75.0
  >=5-point reduction: Week 24: number analyzed (Participants) | 8 | 7
  >=5-point reduction: Week 24 | 62.5 | 71.4
  >=5-point reduction: Week 28: number analyzed (Participants) | 4 | 7
  >=5-point reduction: Week 28 | 100.0 | 85.7
  >=5-point reduction: Week 32: number analyzed (Participants) | 4 | 6
  >=5-point reduction: Week 32 | 50.0 | 100.0
  >=5-point reduction: Week 36: number analyzed (Participants) | 4 | 6
  >=5-point reduction: Week 36 | 75.0 | 83.3
  >=5-point reduction: Week 40: number analyzed (Participants) | 3 | 4
  >=5-point reduction: Week 40 | 100.0 | 50.0
  >=5-point reduction: Week 44: number analyzed (Participants) | 3 | 5
  >=5-point reduction: Week 44 | 100.0 | 60.0
  >=5-point reduction: Week 48: number analyzed (Participants) | 3 | 4
  >=5-point reduction: Week 48 | 100.0 | 75.0
  >=5-point reduction: Week 52: number analyzed (Participants) | 3 | 3
  >=5-point reduction: Week 52 | 100.0 | 66.7
  >=5-point reduction: Week 56: number analyzed (Participants) | 0 | 1
  >=5-point reduction: Week 56 |  | 100.0
  >=5-point reduction: Week 60: number analyzed (Participants) | 0 | 2
  >=5-point reduction: Week 60 |  | 100.0
  >=5-point reduction: Week 64: number analyzed (Participants) | 0 | 1
  >=5-point reduction: Week 64 |  | 100.0
  >=8-point reduction: Week 2 | 16.7 | 15.4
  >=8-point reduction: Week 4: number analyzed (Participants) | 11 | 13
  >=8-point reduction: Week 4 | 27.3 | 30.8
  >=8-point reduction: Week 8: number analyzed (Participants) | 10 | 13
  >=8-point reduction: Week 8 | 40.0 | 30.8
  >=8-point reduction: Week 12: number analyzed (Participants) | 10 | 13
  >=8-point reduction: Week 12 | 40.0 | 30.8
  >=8-point reduction: Week 14: number analyzed (Participants) | 4 | 6
  >=8-point reduction: Week 14 | 25.0 | 16.7
  >=8-point reduction: Week 16: number analyzed (Participants) | 10 | 10
  >=8-point reduction: Week 16 | 60.0 | 40.0
  >=8-point reduction: Week 20: number analyzed (Participants) | 9 | 8
  >=8-point reduction: Week 20 | 55.6 | 62.5
  >=8-point reduction: Week 24: number analyzed (Participants) | 8 | 7
  >=8-point reduction: Week 24 | 50.0 | 57.1
  >=8-point reduction: Week 28: number analyzed (Participants) | 4 | 7
  >=8-point reduction: Week 28 | 100.0 | 57.1
  >=8-point reduction: Week 32: number analyzed (Participants) | 4 | 6
  >=8-point reduction: Week 32 | 50.0 | 66.7
  >=8-point reduction: Week 36: number analyzed (Participants) | 4 | 6
  >=8-point reduction: Week 36 | 75.0 | 33.3
  >=8-point reduction: Week 40: number analyzed (Participants) | 3 | 4
  >=8-point reduction: Week 40 | 100.0 | 50.0
  >=8-point reduction: Week 44: number analyzed (Participants) | 3 | 5
  >=8-point reduction: Week 44 | 100.0 | 60.0
  >=8-point reduction: Week 48: number analyzed (Participants) | 3 | 4
  >=8-point reduction: Week 48 | 100.0 | 75.0
  >=8-point reduction: Week 52: number analyzed (Participants) | 3 | 3
  >=8-point reduction: Week 52 | 66.7 | 66.7
  >=8-point reduction: Week 56: number analyzed (Participants) | 0 | 1
  >=8-point reduction: Week 56 |  | 100.0
  >=8-point reduction: Week 60: number analyzed (Participants) | 0 | 2
  >=8-point reduction: Week 60 |  | 50.0
  >=8-point reduction: Week 64: number analyzed (Participants) | 0 | 1
  >=8-point reduction: Week 64 |  | 100.0

5. Secondary Outcome: Percentage of Participants With Below 8 Points in PRO2
Description: The PRO2 scale is a patient-reported outcome measure specifically used to assess the severity of Crohn's disease. It is derived from the CDAI and focuses on two main symptoms: abdominal pain and stool frequency. Participants rate their abdominal pain on a scale from 0 (none) to 3 (severe) and report the number of soft or liquid stools they have per day, which are then multiplied by a factor of 2 and 5, respectively. The scores from these two components are combined to give an overall PRO2 score ranging from 0 to no upper limit, with a higher score=worse outcome.
Time Frame: At Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percentage of participants
  PRO2 <8 points: Week 2 | 8.3 | 7.7
  PRO2 <8 points: Week 4: number analyzed (Participants) | 11 | 13
  PRO2 <8 points: Week 4 | 9.1 | 7.7
  PRO2 <8 points: Week 8: number analyzed (Participants) | 10 | 13
  PRO2 <8 points: Week 8 | 20.0 | 23.1
  PRO2 <8 points: Week 12: number analyzed (Participants) | 10 | 13
  PRO2 <8 points: Week 12 | 10.0 | 15.4
  PRO2 <8 points: Week 14: number analyzed (Participants) | 4 | 6
  PRO2 <8 points: Week 14 | 0.0 | 16.7
  PRO2 <8 points: Week 16: number analyzed (Participants) | 10 | 10
  PRO2 <8 points: Week 16 | 10.0 | 30.0
  PRO2 <8 points: Week 20: number analyzed (Participants) | 9 | 8
  PRO2 <8 points: Week 20 | 0.0 | 37.5
  PRO2 <8 points: Week 24: number analyzed (Participants) | 8 | 7
  PRO2 <8 points: Week 24 | 12.5 | 28.6
  PRO2 <8 points: Week 28: number analyzed (Participants) | 4 | 7
  PRO2 <8 points: Week 28 | 25.0 | 14.3
  PRO2 <8 points: Week 32: number analyzed (Participants) | 4 | 6
  PRO2 <8 points: Week 32 | 25.0 | 33.3
  PRO2 <8 points: Week 36: number analyzed (Participants) | 4 | 6
  PRO2 <8 points: Week 36 | 0.0 | 16.7
  PRO2 <8 points: Week 40: number analyzed (Participants) | 3 | 4
  PRO2 <8 points: Week 40 | 33.3 | 25.0
  PRO2 <8 points: Week 44: number analyzed (Participants) | 3 | 5
  PRO2 <8 points: Week 44 | 0.0 | 40.0
  PRO2 <8 points: Week 48: number analyzed (Participants) | 3 | 4
  PRO2 <8 points: Week 48 | 0.0 | 50.0
  PRO2 <8 points: Week 52: number analyzed (Participants) | 3 | 3
  PRO2 <8 points: Week 52 | 33.3 | 66.7
  PRO2 <8 points: Week 56: number analyzed (Participants) | 0 | 1
  PRO2 <8 points: Week 56 |  | 100.0
  PRO2 <8 points: Week 60: number analyzed (Participants) | 0 | 2
  PRO2 <8 points: Week 60 |  | 50.0
  PRO2 <8 points: Week 64: number analyzed (Participants) | 0 | 1
  PRO2 <8 points: Week 64 |  | 100.0

6. Secondary Outcome: Percentage of Participants With at Least 50 Percent (%) Improvement in (Endoscopic Response) Simple Endoscopic Score for Crohn's Disease (SES-CD) Score at Week 12
Description: Endoscopic response was defined as a improvement in SES-CD of at least 50% from baseline. The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 (none/unaffected) to 3 (worst). In the SES-CD, each of these 4 components are assessed in the five segments: terminal ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater severity of disease.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percentage of participants | 8.3 [0.2 to 38.5] | 15.4 [1.9 to 45.4]
Statistical Analysis 1: Comparison: E6011 10 mg/kg vs Placebo Then E6011 10 mg/kg; Test type: Superiority; Difference = -7.1, 95% CI 2-sided [-32.1 to 18.0] — The difference of percentage was calculated as E6011 minus placebo

7. Secondary Outcome: Percentage of Participants With Less Than or Equal to (<=) 2 (Endoscopic Remission) SES-CD Score at Week 12
Description: Endoscopic remission was defined as 2 or less points on SES-CD. The SES-CD assesses following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on scale of 0 (none/unaffected) to 3 (worst). In SES-CD, each of these 4 components are assessed in 5 segments: terminal ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater severity of disease.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percentage of participants | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 24.7]
Statistical Analysis 1: Comparison: E6011 10 mg/kg vs Placebo Then E6011 10 mg/kg; Test type: Superiority; Difference = 8.3, 95% CI 2-sided [-7.3 to 24.0] — The difference of percentage was calculated as E6011 minus placebo

8. Secondary Outcome: Change From Baseline in CDAI Score
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. The sub scores of abdominal pain (0-3), general well-being (0-4, higher values mean worse well-being), and number of very soft or liquid stools were then summed. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: Baseline, at Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: FAS was used for analysis. Here "n" = participants who were evaluable for outcome measure at given time points. As planned, combined data for all the periods (remission-induction, rescue and extension periods) was collected and reported in outcome measure due to same dosing of E6011. From Week 14-24, participants data analyzed simultaneously for rescue and extension period and reported collectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
score on a scale
  Change at Week 2 | -38.0 (96.1) | -50.3 (56.7)
  Change at Week 4: number analyzed (Participants) | 11 | 13
  Change at Week 4 | -60.5 (102.7) | -64.5 (91.0)
  Change at Week 8: number analyzed (Participants) | 10 | 13
  Change at Week 8 | -92.8 (109.8) | -70.5 (113.3)
  Change at Week 12: number analyzed (Participants) | 10 | 13
  Change at Week 12 | -92.4 (109.0) | -69.6 (107.0)
  Change at Week 14: number analyzed (Participants) | 4 | 6
  Change at Week 14 | -22.0 (78.1) | -25.8 (100.8)
  Change at Week 16: number analyzed (Participants) | 9 | 9
  Change at Week 16 | -102.8 (95.2) | -89.3 (120.1)
  Change at Week 20: number analyzed (Participants) | 9 | 7
  Change at Week 20 | -115.4 (66.1) | -119.1 (136.4)
  Change at Week 24: number analyzed (Participants) | 8 | 7
  Change at Week 24 | -115.5 (90.1) | -100.0 (120.3)
  Change at Week 28: number analyzed (Participants) | 3 | 7
  Change at Week 28 | -160.7 (28.1) | -153.1 (93.5)
  Change at Week 32: number analyzed (Participants) | 4 | 6
  Change at Week 32 | -97.3 (95.1) | -183.7 (79.1)
  Change at Week 36: number analyzed (Participants) | 4 | 6
  Change at Week 36 | -136.0 (44.2) | -143.0 (109.8)
  Change at Week 40: number analyzed (Participants) | 3 | 4
  Change at Week 40 | -173.7 (49.0) | -157.0 (84.0)
  Change at Week 44: number analyzed (Participants) | 3 | 5
  Change at Week 44 | -147.3 (75.8) | -185.2 (102.9)
  Change at Week 48: number analyzed (Participants) | 3 | 4
  Change at Week 48 | -127.3 (56.1) | -209.8 (99.2)
  Change at Week 52: number analyzed (Participants) | 3 | 3
  Change at Week 52 | -103.7 (102.8) | -171.3 (162.4)
  Change at Week 56: number analyzed (Participants) | 0 | 1
  Change at Week 56 |  | -211.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Change at Week 60: number analyzed (Participants) | 0 | 2
  Change at Week 60 |  | -145.0 (97.6)
  Change at Week 64: number analyzed (Participants) | 0 | 1
  Change at Week 64 |  | -240.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

9. Secondary Outcome: Percent Change From Baseline in CDAI Score
Description: as for outcome 8
Time Frame: Baseline, at Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percent change
  Percent Change at Week 2 | -8.9 (24.6) | -16.7 (21.1)
  Percent Change at Week 4: number analyzed (Participants) | 11 | 13
  Percent Change at Week 4 | -16.0 (26.1) | -20.6 (26.6)
  Percent Change at Week 8: number analyzed (Participants) | 10 | 13
  Percent Change at Week 8 | -25.8 (27.7) | -23.1 (37.1)
  Percent Change at Week 12: number analyzed (Participants) | 10 | 13
  Percent Change at Week 12 | -25.3 (27.1) | -21.8 (33.9)
  Percent Change at Week 14: number analyzed (Participants) | 4 | 6
  Percent Change at Week 14 | -8.3 (28.4) | -9.3 (36.6)
  Percent Change at Week 16: number analyzed (Participants) | 9 | 9
  Percent Change at Week 16 | -29.3 (23.6) | -27.5 (37.0)
  Percent Change at Week 20: number analyzed (Participants) | 9 | 7
  Percent Change at Week 20 | -34.5 (17.5) | -36.6 (45.4)
  Percent Change at Week 24: number analyzed (Participants) | 8 | 7
  Percent Change at Week 24 | -34.8 (25.3) | -32.6 (44.1)
  Percent Change at Week 28: number analyzed (Participants) | 3 | 7
  Percent Change at Week 28 | -53.6 (3.4) | -48.3 (26.2)
  Percent Change at Week 32: number analyzed (Participants) | 4 | 6
  Percent Change at Week 32 | -31.4 (29.3) | -60.1 (28.3)
  Percent Change at Week 36: number analyzed (Participants) | 4 | 6
  Percent Change at Week 36 | -43.3 (10.3) | -43.5 (30.2)
  Percent Change at Week 40: number analyzed (Participants) | 3 | 4
  Percent Change at Week 40 | -53.9 (15.7) | -50.2 (23.7)
  Percent Change at Week 44: number analyzed (Participants) | 3 | 5
  Percent Change at Week 44 | -45.7 (23.1) | -56.8 (27.1)
  Percent Change at Week 48: number analyzed (Participants) | 3 | 4
  Percent Change at Week 48 | -39.6 (17.8) | -63.7 (25.5)
  Percent Change at Week 52: number analyzed (Participants) | 3 | 3
  Percent Change at Week 52 | -33.0 (32.4) | -53.8 (48.2)
  Percent Change at Week 56: number analyzed (Participants) | 0 | 1
  Percent Change at Week 56 |  | -77.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Percent Change at Week 60: number analyzed (Participants) | 0 | 2
  Percent Change at Week 60 |  | -51.9 (37.1)
  Percent Change at Week 64: number analyzed (Participants) | 0 | 1
  Percent Change at Week 64 |  | -87.6 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

10. Secondary Outcome: Change From Baseline in PRO2
Description: as for outcome 5
Time Frame: Baseline, at Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
score on a scale
  Change at Week 2 | -3.1 (6.5) | -4.3 (4.0)
  Change at Week 4: number analyzed (Participants) | 11 | 13
  Change at Week 4 | -5.3 (6.6) | -4.9 (6.5)
  Change at Week 8: number analyzed (Participants) | 10 | 13
  Change at Week 8 | -6.9 (7.3) | -5.8 (7.1)
  Change at Week 12: number analyzed (Participants) | 10 | 13
  Change at Week 12 | -6.5 (6.2) | -5.5 (6.7)
  Change at Week 14: number analyzed (Participants) | 4 | 6
  Change at Week 14 | -3.0 (6.7) | -2.7 (5.4)
  Change at Week 16: number analyzed (Participants) | 10 | 9
  Change at Week 16 | -8.1 (5.7) | -6.1 (7.6)
  Change at Week 20: number analyzed (Participants) | 9 | 7
  Change at Week 20 | -7.9 (4.2) | -8.3 (9.2)
  Change at Week 24: number analyzed (Participants) | 8 | 7
  Change at Week 24 | -6.5 (6.4) | -6.9 (7.4)
  Change at Week 28: number analyzed (Participants) | 3 | 7
  Change at Week 28 | -9.0 (1.0) | -9.6 (5.7)
  Change at Week 32: number analyzed (Participants) | 4 | 6
  Change at Week 32 | -5.5 (6.1) | -12.0 (6.2)
  Change at Week 36: number analyzed (Participants) | 4 | 6
  Change at Week 36 | -9.0 (7.0) | -9.0 (6.1)
  Change at Week 40: number analyzed (Participants) | 3 | 4
  Change at Week 40 | -13.0 (1.7) | -6.3 (6.8)
  Change at Week 44: number analyzed (Participants) | 3 | 5
  Change at Week 44 | -11.0 (2.0) | -9.4 (7.7)
  Change at Week 48: number analyzed (Participants) | 3 | 4
  Change at Week 48 | -8.7 (0.6) | -11.8 (6.6)
  Change at Week 52: number analyzed (Participants) | 3 | 3
  Change at Week 52 | -8.3 (3.1) | -11.0 (8.5)
  Change at Week 56: number analyzed (Participants) | 0 | 1
  Change at Week 56 |  | -13.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Change at Week 60: number analyzed (Participants) | 0 | 2
  Change at Week 60 |  | -9.5 (6.4)
  Change at Week 64: number analyzed (Participants) | 0 | 1
  Change at Week 64 |  | -15.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

11. Secondary Outcome: Percent Change From Baseline in PRO2
Description: as for outcome 5
Time Frame: At Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 12 | 13
percent change
  Percent Change at Week 2 | -13.5 (31.3) | -20.9 (20.0)
  Percent Change at Week 4: number analyzed (Participants) | 11 | 13
  Percent Change at Week 4 | -23.0 (29.8) | -22.9 (28.4)
  Percent Change at Week 8: number analyzed (Participants) | 10 | 13
  Percent Change at Week 8 | -30.1 (33.0) | -29.2 (34.6)
  Percent Change at Week 12: number analyzed (Participants) | 10 | 13
  Percent Change at Week 12 | -29.4 (28.0) | -25.8 (31.0)
  Percent Change at Week 14: number analyzed (Participants) | 4 | 6
  Percent Change at Week 14 | -13.4 (28.6) | -17.6 (32.7)
  Percent Change at Week 16: number analyzed (Participants) | 10 | 9
  Percent Change at Week 16 | -36.8 (25.0) | -27.9 (34.4)
  Percent Change at Week 20: number analyzed (Participants) | 9 | 7
  Percent Change at Week 20 | -36.2 (16.8) | -37.6 (46.7)
  Percent Change at Week 24: number analyzed (Participants) | 8 | 7
  Percent Change at Week 24 | -30.0 (28.0) | -35.9 (41.1)
  Percent Change at Week 28: number analyzed (Participants) | 3 | 7
  Percent Change at Week 28 | -47.7 (9.2) | -46.2 (23.7)
  Percent Change at Week 32: number analyzed (Participants) | 4 | 6
  Percent Change at Week 32 | -25.1 (32.7) | -58.3 (30.3)
  Percent Change at Week 36: number analyzed (Participants) | 4 | 6
  Percent Change at Week 36 | -37.1 (25.5) | -42.9 (24.6)
  Percent Change at Week 40: number analyzed (Participants) | 3 | 4
  Percent Change at Week 40 | -56.4 (14.3) | -31.2 (32.6)
  Percent Change at Week 44: number analyzed (Participants) | 3 | 5
  Percent Change at Week 44 | -46.9 (9.1) | -45.3 (32.5)
  Percent Change at Week 48: number analyzed (Participants) | 3 | 4
  Percent Change at Week 48 | -37.3 (7.2) | -57.2 (26.7)
  Percent Change at Week 52: number analyzed (Participants) | 3 | 3
  Percent Change at Week 52 | -38.4 (22.2) | -56.1 (34.6)
  Percent Change at Week 56: number analyzed (Participants) | 0 | 1
  Percent Change at Week 56 |  | -81.3 (NA) — Standard deviation could not be estimated due to insufficient number of participants.
  Percent Change at Week 60: number analyzed (Participants) | 0 | 2
  Percent Change at Week 60 |  | -59.4 (39.8)
  Percent Change at Week 64: number analyzed (Participants) | 0 | 1
  Percent Change at Week 64 |  | -93.8 (NA) — Standard deviation could not be estimated due to insufficient number of participants.

12. Secondary Outcome: Change From Baseline in SES-CD Score at Week 12
Description: The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 (none/unaffected) to 3 (worst). In the SES-CD, each of these 4 components are assessed in the five segments: terminal ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater severity of disease.
Time Frame: Baseline, at Week 12
Population: FAS was used for analysis. Here, "overall number of participants analyzed" ('N') = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 10 | 13
score on a scale | 1.4 (4.9) | -3.5 (4.9)

13. Secondary Outcome: Percent Change From Baseline in SES-CD Score at Week 12
Description: as for outcome 12
Time Frame: Baseline, at Week 12
Population: FAS was used for analysis. Here "overall number of participants analyzed" ('N') = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 10 | 13
percent change | -0.3 (45.6) | -19.2 (33.2)

14. Secondary Outcome: Percentage of Participants Who Achieved Steroid-free Remission up to Week 64
Description: Steroid-free remission was defined as clinical remission (CDAI remission or PRO2-remission) in participants who became steroid free through steroid reduction. CDAI remission was defined as CDAI score below 150 points. PRO2-remission was defined as PRO2- score less than 8-points. The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. The total CDAI score ranged from 0-600 with a higher score indicating a worse outcome. Participants for PRO2 scale rate their abdominal pain on scale from 0 (none) to 3 (severe) and report the number of soft or liquid stools they have per day, which are then multiplied by a factor of 2 and 5, respectively. Scores from two components combined to give overall score ranging from 0 to no upper limit, with higher score=worse outcome.
Time Frame: Up to Week 64
Population: FAS was used for analysis. Here, "overall number of participants analyzed" ('N') = participants who were evaluable for this outcome measure. As planned, combined data for all the periods (remission-induction, rescue and extension periods) was collected and reported in outcome measure due to same dosing of E6011. Steroid-free remission was assessed in participants who were concomitantly taking adrenocorticosteroid.
Measure: Number; unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 3 | 6
percentage of participants | 0 | 0

15. Secondary Outcome: Percentage of Participants Who Achieved Steroid-free Improvement up to Week 64
Description: Steroid-free clinical improvement = clinical response (CR70 response, CR100 response, PRO2-CR5 and PRO2-CR8 responses) in participants who became steroid free through steroid reduction. CR70 and CR100 = clinical response with decrease of >=70 point and >=100 point from baseline, respectively in CDAI. PRO2-CR5 and PRO2-CR8 = clinical response with decrease of >=5 point and >=8 point from baseline, respectively in PRO2. CDAI system was composite index of 8 disease activity variables. Total CDAI score ranged 0-600; higher score = worse outcome. Participants for PRO2 scale rate their abdominal pain on scale from 0 (none) to 3 (severe); report number of soft or liquid stools they have per day, which are multiplied by factor of 2 and 5, respectively. The scores from these two components are combined to give an overall PRO2 score ranging from 0 to no upper limit, with a higher score=worse outcome.
Time Frame: Up to Week 64
Population: FAS was used for analysis. Here, "overall number of participants analyzed" ('N') = participants who were evaluable for this outcome measure. As planned, combined data for all the periods (remission-induction, rescue and extension periods) was collected and reported in outcome measure due to same dosing of E6011. Steroid-free improvement was assessed in participants who were concomitantly taking adrenocorticosteroid.
Measure: Number; unit: percentage of participants
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 3 | 6
percentage of participants | 0 | 0

16. Secondary Outcome: Change From Baseline in Steroid Dosage in Participants Concomitantly Using Adrenocorticosteroids up to Week 64
Description: Change from baseline in steroid dosage in participants concomitantly using adrenocorticosteroids up to Week 64 was reported.
Time Frame: Baseline up to Week 64
Population: FAS was used for analysis. Here, "N" = participants who were evaluable for this outcome measure. As planned, combined data for all the periods (remission-induction, rescue, extension and post observation periods) was collected and reported in outcome measure due to same dosing of E6011.
Measure: Mean (Standard Deviation); unit: milligram per day (mg/day)
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 3 | 6
milligram per day (mg/day) | 0 (0) | 0 (0)

17. Secondary Outcome: Percent Change From Baseline in Steroid Dosage in Participants Concomitantly Using Adrenocorticosteroids up to Week 64
Description: Percent change from baseline in steroid dosage in participants concomitantly using adrenocorticosteroids up to Week 64 was reported.
Time Frame: Baseline up to Week 64
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E6011 10 mg/kg | Placebo Then E6011 10 mg/kg
Number analyzed (Participants) | 3 | 6
percent change | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Remission induction period: From the first dose of the study drug (Week 0) up to Week 12; Rescue period: From Week 12 up to Week 24; Extension period: Week 12 up to Week 64; Post-observation period: Up to 70 days after last dose of study drug
Groups:
- Remission Induction Period: E6011 10 mg/kg: Participants received E6011 10 mg/kg, IV infusion once, at Weeks 0,1, 2 then every 2 weeks up Week 10 during Remission Induction Period.
- Remission Induction Period: Placebo: Participants received placebo, IV infusion once, at Weeks 0,1, 2 then every 2 weeks up Week 10 during Remission Induction Period.
- Rescue Period: E6011 10 mg/kg: Participants received E6011 10 mg/kg, IV infusion once, at Weeks 12, 13, 14 then every 2 weeks up to Week 22 during Rescue Period.
- Rescue Period: Placebo to E6011 10 mg/kg: Participants who received placebo in the remission induction period received E6011 10 mg/kg, IV infusion once, at Weeks 12, 13, 14 then every 2 weeks up to Week 22 during Rescue the Period.
- Extension Period: E6011 10 mg/kg: Participants with response at Week 12 and Week 24 received E6011 10 mg/kg, IV infusion once, every 4 weeks from Week 12 to Week 48 and Week 24 to Week 60, respectively, during the Extension Period.
- Extension Period: Placebo to E6011 10 mg/kg: Participants who received placebo in the remission induction period, who had response at Week 12 and Week 24 received E6011 10 mg/kg, IV infusion once, every 4 weeks from Week 12 to Week 48 and Week 24 to Week 60, respectively during the Extension Period.
- Post-observation Period: E6011 10 mg/kg: Participants who received E6011 10 mg/kg in any of the treatment periods were observed during Post-observation Period for 70 days after last dose.
- Post-observation Period: Placebo to E6011 10 mg/kg: Participants who received placebo in the remission induction period and who were switched to receive E6011 10 mg/kg in Rescue or Extension periods were observed during Post-observation Period for 70 days after last dose.
Arm/Group | Remission Induction Period: E6011 10 mg/kg | Remission Induction Period: Placebo | Rescue Period: E6011 10 mg/kg | Rescue Period: Placebo to E6011 10 mg/kg | Extension Period: E6011 10 mg/kg | Extension Period: Placebo to E6011 10 mg/kg | Post-observation Period: E6011 10 mg/kg | Post-observation Period: Placebo to E6011 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/5 | 0/7 | 0/7 | 0/8 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/13 | 0/5 | 2/7 | 0/7 | 0/8 | 0/12 | 1/13
Other Adverse Events (participants affected / at risk) | 6/12 | 5/13 | 3/5 | 4/7 | 1/7 | 5/8 | 2/12 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remission Induction Period: E6011 10 mg/kg (N=12) | Remission Induction Period: Placebo (N=13) | Rescue Period: E6011 10 mg/kg (N=5) | Rescue Period: Placebo to E6011 10 mg/kg (N=7) | Extension Period: E6011 10 mg/kg (N=7) | Extension Period: Placebo to E6011 10 mg/kg (N=8) | Post-observation Period: E6011 10 mg/kg (N=12) | Post-observation Period: Placebo to E6011 10 mg/kg (N=13)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remission Induction Period: E6011 10 mg/kg (N=12) | Remission Induction Period: Placebo (N=13) | Rescue Period: E6011 10 mg/kg (N=5) | Rescue Period: Placebo to E6011 10 mg/kg (N=7) | Extension Period: E6011 10 mg/kg (N=7) | Extension Period: Placebo to E6011 10 mg/kg (N=8) | Post-observation Period: E6011 10 mg/kg (N=12) | Post-observation Period: Placebo to E6011 10 mg/kg (N=13)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT03733314/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT03733314/SAP_001.pdf